CLINICAL TRIAL: NCT05145907
Title: A Multicenter, Open-label, Exploratory Phase II Clinical Study to Evaluate the Safety and Tolerability and Preliminary Efficacy of TJ107 Combine With Pembrolizumab Injection in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study to Evaluate Safety and Efficacy of TJ107 Combine With PD-1 in Patients With Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ107001STM202
Record Dates: First submitted 2021-11-01; First posted 2021-12-06 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Triple-negative Breast Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: Triple-negative breast cancer; Head and neck squamous cell carcinoma; Solid Tumors
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Open-label, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJ107+Pembrolizumab (Experimental): TJ107 1200ug/Kg,Q12W + Pembrolizumab 200mg Q3W
  Interventions: Biological: TJ107 +Pembrolizumab

INTERVENTIONS:
Biological: TJ107 +Pembrolizumab — TJ107 injection:1200ug/Kg, Q12W, IM; Pembrolizumab: 200mg, Q3W, IV

SUMMARY:
Study Purpose and Design:A Multicenter, Open-label, Exploratory Phase II Clinical Study to Evaluate the Safety and Tolerability and Preliminary Efficacy of TJ107 in Combination with Pembrolizumab Injection in Patients with Locally Advanced or Metastatic Solid Tumors

DETAILED DESCRIPTION:
This open-label, multicenter phase 2 study will enroll 28 to 39 subjects in each of the following 4 cohorts Cohort 1 Triple-negative breast cancer Cohort 2 Head and neck squamous cell carcinoma Cohort 3 Other tumor species (to be determined) Cohort 4 Other tumor species (to be determined) The trial consists of two phases, the first is a safety run-in phase and the second is a case extension phase.

In the safety run-in phase, 3 subjects will be treated with TJ107 (1200 µg/kg q12w) combined with Pembrolizumab Injection (200 mg q3w) first. A safety assessment was conducted by a safety assessment committee composed of the sponsor and the investigator on the first dose in these 3 subjects to determine that the dose of TJ107 1200 µg/kg was safe and to determine whether to continue the safety assessment in these 3 patients, either at this dose level, or at a dose or dosing interval adjustment (e.g., the dose of TJ107 was adjusted to 960 ug/kg or the dosing interval was adjusted).

In the case expansion phase, 28-39 subjects will be enrolled in each cohort, and TJ107 (1200 µg/kg q12w) combined with Pembrolizumab Injection (200 mg q3w) or TJ107 adjusted dose combined with Pembrolizumab Injection (200 mg q3w) will be administered until intolerance or disease progression and other endpoint events occur.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged over 18 years (inclusive);
* ECOG score: 0 - 2 points
* Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors, including TNBC and HNSCC
* No previous treatment with CPI
* Agreement to provide a previously archived tumor tissue specimen or biopsy to collect tumor lesion tissue
* Subject has at least 1 measurable lesion as defined by RECIST V1.1
* Expected survival ≥ 6 months
* Adequate organ function
* Males of childbearing potential or females of childbearing potential must use highly effective contraceptive methods during the trial and continuing for 6 months after the last dose
* The subject voluntarily joined the study and signed an informed consent form

Exclusion Criteria:

* Pregnant or lactating women;
* Prior cell therapy;
* Received systemic anti-tumor therapy within 2 weeks or 5 half-lives of the treatment agent (whichever is shorter) before the start of treatment;
* Previous or current presence of two or more primary tumors
* Patients with active autoimmune diseases
* Have received systemic treatment with corticosteroids (10 mg prednisone equivalent daily) or other immunosuppressive agents for more than 7 days within 2 weeks before the start of treatment
* Received investigational drugs within 2 weeks before the start of treatment;
* Major surgery or serious trauma within 4 weeks before the start of treatment;
* Patients with symptomatic central nervous system (CNS) metastasis
* Active viral infectious disease requiring systemic treatment at screening:
* Known serious hypersensitivity history
* Uncontrolled pleural effusion, ascites, or pericardial effusion at screening;
* Presence or history of active interstitial lung disease;
* Patients with hypertension that cannot be well controlled with medical therapy.
* Presence of clinically significant cardiovascular disease
* Deep venous thrombosis within 6 months before the start of treatment
* Thrombolytic therapy within 10 days prior to the start of treatment
* Any active infection requiring intravenous anti-infective therapy before the start of treatment
* Had toxicity not resolved to ≤ Grade 1 (CTCAE 5.0) from previous anticancer therapy
* Known or suspected inability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of Adverse events | Through the study assessed up to 2 years
  The rate of Adverse events
The rate of Senior Adverse Events | Through the study assessed up to 2 years
  The rate of Senior Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Liyang Song, Master, Study Director — I-Mab Biopharma US Limited
Locations (20):
- China (20):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangzhou
  - Hainan General Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of Huzhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jilin Guowen Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Yanbian University Hospital, Yanji, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital,Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No